CLINICAL TRIAL: NCT03961724
Title: Combination of Neuroimaging and Metabolomics of Brain Impairment in Patients With End-stage Renal Disease: a Multi-center Prospective Cohort Study
Brief Title: Neuroimaging and End Stage Renal Disease
Acronym: NESRD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: 215 Hospital of Shaanxi NI (Other); Baoji Zhongxin Hospital (Unknown); Taihe Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2018-006
Record Dates: First submitted 2019-04-26; First posted 2019-05-23 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESRD group
  Interventions: Device: magnetic resonance image (MRI)
- Control group
  Interventions: Device: magnetic resonance image (MRI)

INTERVENTIONS:
Device: magnetic resonance image (MRI) — serum metabolomics
  Other Names: serum

SUMMARY:
Brain impairment is one of the common complications of end-stage renal disease (ESRD). The patients always present with various cerebrovascular diseases, cognitive impairment and sensorimotor abnormalities, with morbidity over 40%. However, the risk factors and the neural mechanisms of brain injury in ESRD is still unclear. Identifying the risk factors and finding objective and reliable biomarkers of brain impairment in the process of ESRD is an important clinical problem. At the same time, to find the neural mechanisms of brain damage in ESRD is a serious scientific problem. Neuroimaging techniques based on multi-modal magnetic resonance image (MRI) can detect the structural and functional brain abnormalities objectively and sensitively, especially for those without obvious clinical symptoms. Through the deep analysis of brain MRI data, it is helpful for studying the neural mechanisms of brain damage in ESRD in the perspective from brain science. In addition, the accumulation of uremic toxins is supposed to play an essential role in the brain impairment of ESRD. The metabolomics is a useful method in detecting the uremic toxins with different molecular weights. In this study, the investigators will collect the brain MRI, serum metabolomics and cognitive assessment data before the dialysis initiation, and then will make prospective longitudinal observation of changes of brain impairment during the dialysis. Thus, combining analysis of neuroimaging and metabolomics will provide more information for finding the risk factors and imaging diagnostic markers of brain impairment in ESRD. It will also helpful for explaining the underlying mechanisms of brain impairment in ESRD, providing an objective basis for clinical diagnosis and prediction of the prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with end stage renal disease before dialysis initiation
* Chronic renal failure
* Chronic renal failure
* 18-55 years old
* Right handedness

Exclusion Criteria:

* Concurrent severe infection
* With other severe diseases
* History of central nervous system diseases, such as mental disorder, degenerative diseases of central nervous system, tumors, trauma, etc.
* History of alcohol dependence and drug abuse
* History of brain operation
* Loss of vision or hearing
* Psychotropic medication in three months
* Contraindication of MRI examination, such as metal implants and claustrophobia, and other reasons that cannot cooperate with MRI examination
* Cerebrovascular diseases which can be detected from conventional MR images, including the size of cerebral hemorrhage over 10 mm, infarction over 20 mm, subarachnoid hemorrhage, subdural hemorrhage and extradural hemorrhage.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All of the patients of ESRD group are in-patients and out-patients in the nephrology department from three research centers. The subjects of control group are recruited from community.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline brain structure measures at 3 months and 12months | baseline (before dialysis initiation), hemodialysis for 3 months and 12 months
  The changes of brain volume (mm3) are evaluated by structural MRI
Change from baseline brain function measures at 3 months and 12months | baseline (before dialysis initiation), hemodialysis for 3 months and 12 months
  The changes of brain functional connectivity intensity are evaluated by functional MRI

SECONDARY OUTCOMES:
Changes from baseline cognitive condition at 3 months and 12months | baseline (before dialysis initiation), hemodialysis for 3 months and 12 months
  The cognitive condition is assessed by Montreal cognitive assessment (MoCA). The MoCA assesses several cognitive domains: 1) visuospatial and executive abilities are assessed using a trail-making test B (1 point), clock-drawing task (3 points) and a cube copy (1 point); 2) naming is assessed with low-familiarity animals (3 points); 3) the short-term memory (5 points) involves two learning trials of five nouns; 4) attention are evaluated using a sustained attention task (1 point), a serial subtraction task (3 points), and digits forward and backward (1 point each); 5) language is assessed using a repetition of two syntactically complex sentences (2 points), and the verbal fluency task (1 point); 6) orientation to time and place is evaluated by asking the subject for the date and the city (6 points). The scale ranges is from 0 to 30, and score of 26 or over is considered to be normal. Subscales are summed to compute a total score, and higher values represent a better outcome.
Changes from baseline depression condition at 3 months and 12months | baseline (before dialysis initiation), hemodialysis for 3 months and 12 months
  The affective complaints are assessed by Beck depression inventory (BDI). The BDI is a 21-question multiple-choice self-report inventory in the past week, for measuring the severity of depression. The BDI is composed of items relating to symptoms of depression such as hopelessness and irritability, cognitions such as guilt or feelings of being punished, as well as physical symptoms such as fatigue, weight loss, and lack of interest in sex. Each question had a set of at least four possible responses, ranging in intensity: (0) I do not feel sad; (1) I feel sad; (2) I am sad all the time and I can't snap out of it; (3) I am so sad or unhappy that I can't stand it. When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is summed to be compared to a key to determine the depression's severity. The scale ranges is from 0 to 63, and the higher total scores indicate more severe depressive symptoms.
Changes from baseline anxiety condition at 3 months and 12months | baseline (before dialysis initiation), hemodialysis for 3 months and 12 months
  The affective complaints are assessed by Beck anxiety inventory (BAI). The BAI is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults. The questions used in this measure ask about common symptoms of anxiety that the subject has had during the past week (including the day you take it) (such as numbness and tingling, sweating not due to heat, and fear of the worst happening). The BAI contains 21 questions, each answer being scored on a scale value of 1 (not at all) ,2 (mild), 3 (moderate), to 4 (severely). The scale ranges is from 21 to 84 , and higher total scores indicate more severe anxiety symptoms.
Changes from baseline serum metabolomics at 3 months and 12months | baseline (before dialysis initiation), hemodialysis for 3 months and 12 months
  The serum metabolomics are conducted by liquid Chromatograph Mass Spectrometer (LC-MS), mainly including the molecules of uremic toxins.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhang, PhD, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu X, Ma S, Liu S, Luo Z, Zhu Q, Yuan H, Zhu X, Gu W, Li P, Zhang J, Zhang M, Mu J. Structural Connectivity Disruption and Structural-Functional Decoupling in Working Memory Networks Across Pre-Dialysis and Maintenance Hemodialysis End-Stage Renal Disease Patients. CNS Neurosci Ther. 2026 Jan;32(1):e70761. doi: 10.1002/cns.70761. PMID 41552885